CLINICAL TRIAL: NCT05111795
Title: Holmium-166 Retrospective Collection of Real-World Data
Acronym: RECORD
Status: Completed | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T141E4
Record Dates: First submitted 2021-10-12; First posted 2021-11-08 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma; Metastatic Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Selective Internal Radiation Therapy with QuiremSpheresTM Holmium-166 Microspheres — SIRT work-up procedure and SIRT procedure
  Other Names: SIRT, Radioembolization, TARE

SUMMARY:
The primary objective of the study is to further describe the general safety and clinical performance of QuiremSpheresTM Holmium-166 Microspheres and QuiremScoutTM Holmium-166 Microspheres in a real-world post-market setting, with specific attention to outcomes per tumor origin.

DETAILED DESCRIPTION:
This study, with an observational retrospective longitudinal design, is intended to collect data from the devices (QuiremScoutTM Holmium-166 Microspheres, QuiremSpheresTM Holmium-166 Microspheres, and where available, Q-SuiteTM) used in a post-market, real-world setting. It is non-comparative due to the retrospective nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of primary liver tumor or metastases in the liver.
* Patients treated with QuiremScoutTM Holmium-166 Microspheres and/or QuiremSpheresTM Holmium-166 Microspheres from 15 July 2019 to 15 July 2021.
* Patient is ≥ 18 years.
* If required by national regulation, patient has understood and signed written informed consent to retrospective data collection.

Exclusion Criteria:

* Patients previously included in prospective interventional study with QuiremScoutTM Holmium-166 Microspheres and/or QuiremSpheresTM Holmium-166 Microspheres.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be included has been treated at the top-ordering hospitals for QuiremSpheresTM Holmium-166 Microspheres. All patients treated at these hospitals between 15 July 2019 and 15 July 2021 are aimed to be included.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events | 30 months
  The primary safety endpoint is defined in terms of incidence of adverse events CTCAE (Common Terminology Criteria for Adverse Events) grade ≥ 3, or any grade of a predefined list of events stemming from risk management of QuiremSpheresTM Holmium-166 Microspheres and QuiremScoutTM Holmium-166 Microspheres.
Progression Free Survival (PFS) | 30 months
  Time from SIRT procedure until overall progression or death
Hepatic Progression Free Survival (HPFS) | 30 months
  Time from SIRT procedure until progression in the liver or death
Overall survival (OS) | 30 months
  Time from SIRT procedure until death from any cause
Tumor response in the liver | 3 months
  Response as per routine practice following the guidelines for corresponding tumor type
Lung shunt prediction | 1 month
  Lung shunt prediction will be evaluated by comparing the predicted and actual lung shunt, either in terms of percentage or absorbed dose

SECONDARY OUTCOMES:
Administered activity | 1 month
  The technical performance of SIRT in term of administered activity in Becquerel (GBq or MBq) with QuiremSpheresTM Holmium-166 Microspheres.
Liver volume treated | 1 month
  The technical performance of SIRT in term of liver volume treated in mL with QuiremSpheresTM Holmium-166 Microspheres.
SIRT treatment approach | 1 month
  The technical performance of SIRT in term of treatment approach (selective, lobar, bi-lobar, whole liver) with QuiremSpheresTM Holmium-166 Microspheres.
Tumor absorbed dose | 1 month
  The technical performance of SIRT in term of tumor absorbed dose in Gray (Gy) recorded from post-treatment imaging or based on injected activity and target volume with QuiremSpheresTM Holmium-166 Microspheres.
Normal liver absorbed dose | 1 month
  The technical performance of SIRT in term of normal liver absorbed dose in Gray (Gy) recorded from post-treatment imaging or based on injected activity and target volume with QuiremSpheresTM Holmium-166 Microspheres.
The use of Q-SuiteTM in clinical practice | 1 month
  The use of Q-SuiteTM in clinical practice will be recorded based on the software which is mentioned in the description of treatment or the presence of a Q-SuiteTM generated report in the patient's medical file.
Number of patients downstaged to liver resection or liver transplantation | 30 months
  The number of patients downstaged to liver resection or liver transplantation will be reviewed based on the number of patients that underwent liver resection or liver transplantation after the SIRT procedure

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (3):
  - ASZ Aalst, Aalst
  - OLV Aalst, Aalst
  - CUB Hôpital Erasme, Brussels
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Klinikum Herford, Herford
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin Rostock, Rostock
- IFO IRCCS - Istituto Nazionale Tumori Regina Elena, Rome, Italy
- University Medical Center Utrecht, Utrecht, Netherlands
- Instituto Português De Oncologia Do Porto Francisco Gentil, EPE, Porto, Portugal
- Hospital Universitari Germans Trias i Pujol, Barcelona, Spain
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No